CLINICAL TRIAL: NCT04747691
Title: Assessing Gastric Motility and Distention in Postoperative Gastrointestinal Surgery Using Bedside Gastric Ultrasound: Predicting Risk of Aspiration Pneumonia, Ileus, Return of Bowel Function
Status: Completed | Type: Observational
Sponsor: Eric Schwenk (Other)
Responsible Party: Sponsor-Investigator, Eric Schwenk, Associate Professor of Anesthesiology and Orthopedic Surgery, Thomas Jefferson University
Organization: Thomas Jefferson University (Other)
Other Study IDs: 20D.1009
Record Dates: First submitted 2021-02-05; First posted 2021-02-10 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-06

CONDITIONS: Postoperative Ileus; Postoperative Nausea; Postoperative Complications; Postoperative Nausea and Vomiting; Postoperative Vomiting; Aspiration Vomitus
Keywords: Postoperative Complications; Postoperative Ileus
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Postoperative Complications; Respiratory Aspiration of Gastric Contents

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients assessed with postoperative bedside gastric ultrasound: This patient population will include postoperative patients who received a gastrointestinal surgery and are being assessed with the bedside gastric ultrasound.
  Interventions: Diagnostic Test: Bedside gastric ultrasound

INTERVENTIONS:
Diagnostic Test: Bedside gastric ultrasound — Bedside ultrasound exam of the stomach

SUMMARY:
Point-of-care gastric ultrasound will be used to measure stomach contents postoperative in patients who underwent colorectal surgery. Stomach volume and status (empty or full) will be compared retrospectively to the standard clinical criteria for diet advancement to determine if stomach volume via ultrasound is associated with successful diet advancement, nausea/vomiting, nasogastric tube replacement, length of stay, and other clinical outcomes. Clinicians performing clinical care will be blinded to the ultrasound exam results.

DETAILED DESCRIPTION:
Patient population: Patients undergoing colorectal surgery will be enrolled prospectively (both cancer and non-cancer patients).

Inclusion Criteria:

* Patients aged > 18 years of age
* Patients undergoing colorectal surgery (both cancer and non-cancer)

Exclusion Criteria:

* Patients < 18 years of age
* Patients with previous gastric surgery

  * Patients with inadequate or difficult baseline gastric ultrasound images
  * Any other patient deemed a poor study candidate by the treating physicians

Research Design/Protocol: We will perform postoperative point-of-care ultrasound examinations in colorectal surgery patients and will record gastric volumes at set time points, including preoperative and the morning of postoperative day 1. The surgical team, who will be blinded to the results of the ultrasound exam, will make decisions to advance diet, remove nasogastric tube, and begin oral medications based on standard clinical criteria. At the completion of the study we will determine if there is any association between gastric volume on ultrasound and patient complications, such as nausea/vomiting, replacement of nasogastric tube, aspiration of gastric contents, inability to tolerate solid diet, prolonged admission/length of stay, and other clinical outcomes.

Outcomes: Our exploratory outcome measures will be tolerance of diet, replacement of NG tube, nausea/vomiting, time to flatus, aspiration pneumonia/pneumonitis, and length of stay.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged > 18 years of age
* Patients undergoing colorectal surgery (both cancer and non-cancer)

Exclusion Criteria:

* Patients < 18 years of age
* Patients with previous gastric surgery

  * Patients with difficult or poor ultrasound images at baseline
  * Any patient deemed a poor candidate by the treating physicians

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients scheduled for colorectal surgery
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Tolerance of diet advancement | 0 - 14 days
  Includes replacement of NGT, downgrading diet

SECONDARY OUTCOMES:
Emesis | 0 - 14 days
Time to first flatus | 0 - 14 days
Aspiration pneumonitis | 0 - 14 days
  Clinical or radiographic evidence of aspiration
Time to first bowel movement | 0 - 14 days

OTHER OUTCOMES:
Nausea | 0 - 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haskins SC, Kruisselbrink R, Boublik J, Wu CL, Perlas A. Gastric Ultrasound for the Regional Anesthesiologist and Pain Specialist. Reg Anesth Pain Med. 2018 Oct;43(7):689-698. doi: 10.1097/AAP.0000000000000846. PMID 30052550
- [Background] Gola W, Domagala M, Cugowski A. Ultrasound assessment of gastric emptying and the risk of aspiration of gastric contents in the perioperative period. Anaesthesiol Intensive Ther. 2018;50(4):297-302. doi: 10.5603/AIT.a2018.0029. Epub 2018 Sep 17. PMID 30221339
- [Background] Mirbagheri N, Dunn G, Naganathan V, Suen M, Gladman MA. Normal Values and Clinical Use of Bedside Sonographic Assessment of Postoperative Gastric Emptying: A Prospective Cohort Study. Dis Colon Rectum. 2016 Aug;59(8):758-65. doi: 10.1097/DCR.0000000000000637. PMID 27384094
- [Background] Sabate S, Mazo V, Canet J. Predicting postoperative pulmonary complications: implications for outcomes and costs. Curr Opin Anaesthesiol. 2014 Apr;27(2):201-9. doi: 10.1097/ACO.0000000000000045. PMID 24419159
- [Background] Warner MA, Warner ME, Weber JG. Clinical significance of pulmonary aspiration during the perioperative period. Anesthesiology. 1993 Jan;78(1):56-62. doi: 10.1097/00000542-199301000-00010. PMID 8424572
- [Background] Zhang X, Zheng W, Chen C, Kang X, Zheng Y, Bao F, Gan S, Zhu S. Goal-directed fluid therapy does not reduce postoperative ileus in gastrointestinal surgery: A meta-analysis of randomized controlled trials. Medicine (Baltimore). 2018 Nov;97(45):e13097. doi: 10.1097/MD.0000000000013097. PMID 30407319
- [Background] Wolthuis AM, Bislenghi G, Fieuws S, de Buck van Overstraeten A, Boeckxstaens G, D'Hoore A. Incidence of prolonged postoperative ileus after colorectal surgery: a systematic review and meta-analysis. Colorectal Dis. 2016 Jan;18(1):O1-9. doi: 10.1111/codi.13210. PMID 26558477
- [Background] Barletta JF, Senagore AJ. Reducing the burden of postoperative ileus: evaluating and implementing an evidence-based strategy. World J Surg. 2014 Aug;38(8):1966-77. doi: 10.1007/s00268-014-2506-2. PMID 24682277
- [Background] Vather R, O'Grady G, Bissett IP, Dinning PG. Postoperative ileus: mechanisms and future directions for research. Clin Exp Pharmacol Physiol. 2014 May;41(5):358-70. doi: 10.1111/1440-1681.12220. PMID 24754527